CLINICAL TRIAL: NCT07020130
Title: Risk Factors,PREvention and outComes for Contrast-Induced Acute Kidney Injury in patientS undErgoing Percutaneous Coronary Intervention：a Single-center Cohort Study(PRECISE)
Brief Title: Risk Factors,PREvention and OutComes for CI-AKI in PatientS undErgoing PCI (PRECISE)
Acronym: PRECISE
Status: Completed | Type: Observational
Sponsor: Kaiyang Lin (Other)
Responsible Party: Sponsor-Investigator, Kaiyang Lin, Director, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: K2019-07-011
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: CIN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study included all patients undergoing percutaneous coronary intervention(PCI) in Fujian Provincial Hospital from January 1st 2012 to December 31st 2018. The aim was to determine the incidence,risk factors,prophylactic strategy and outcomes of CI-AKI in patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients undergoing PCI at ICU

Exclusion Criteria:

* pregnancy lactation end-stage renal disease (eGFR <15 mL/min/1.73 m2) long-term dialysis treatment intravascular administration of contrast medium within the last 7 or 3 days postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Critically ill patients undergoing PCI at ICU were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 3030 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
CI-AKI | 5 year
  This was due to acute kidney injury following the use of intravascular contrast media. Serum creatinine is the primary measuring modalities.
CKD | 5 year
  Chronic renal structural and functional disorders that occurred during follow-up after administration of intravascular contrast agents, estimated glomerular filtration rate (eGFR) as the primary measuring modalities.

SECONDARY OUTCOMES:
all-cause mortality | 5 year
  Defined as deaths occurring during follow-up after discharge from EPCI, excluding force majeure factors such as natural disasters and car accidents,and the necessary information was gathered during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided